CLINICAL TRIAL: NCT04868175
Title: The Effects of Topical Beta Blocker and Prostaglandin on Interval Intraocular Pressure in Intravitreal Injection - a Randomised Controlled Prospective Study
Brief Title: Interval Intraocular Pressure in Intravitreal Injection Study
Acronym: IIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IIII
Record Dates: First submitted 2021-04-20; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Glaucoma; Intraocular Pressure
MeSH Terms: conditions — Glaucoma | interventions — Timolol; Travoprost; Hypromellose Derivatives

STUDY DESIGN:
Intervention Model Description: Group 1: control (hypromellose), then Timolol, then Travatan Group 2: Timolol, then Travatan, Hypromellose Group 3: Travatan, then Hypromellose, Timolol
  There are three groups of different treatments. Patients recruited will undergone all three groups of treatments. During the first injection visit, patients will be randomized (by envelope method upon recruitment) to start with one of the three groups by envelope method. Treatment given to each group according to randomization in the first visit, then rotated to second and third group at two subsequent injections accordingly.
  Injection doctors masked to treatments given.
Who Masked: Participant, Care Provider
Masking Description: Patients are not exposed to the eye drop bottle (taped) and the doctors measuring pressure and performing the intravitreal injections are not shown the eye drops given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): control (hypromellose), then Timolol, then Travatan
  Interventions: Drug: Timolol; Drug: Travatan; Drug: Hypromellose
- Group 2 (Active Comparator): Timolol, then Travatan, Hypromellose
  Interventions: Drug: Timolol; Drug: Travatan; Drug: Hypromellose
- Group 3 (Active Comparator): Travatan, then Hypromellose, Timolol
  Interventions: Drug: Timolol; Drug: Travatan; Drug: Hypromellose

INTERVENTIONS:
Drug: Timolol — Topical eye drops for lowering intraocular pressure Beta blocker to reduce aqueous production
Drug: Travatan — Topical eye drops for lowering intraocular pressure Prostaglandin analogue to increase aqueous outflow
Drug: Hypromellose — Placebo eye drop, lubricant

SUMMARY:
This is a prospective study of IOP in Intravitreal injections to evaluate:

1. IOP effect of intravitreal injection
2. IOP response to prophylactic beta blocker or Prostaglandin vs control (Hypromellose) over multiple time periods
3. IOP response in correlation to number of injections, IOL, type of anti VEGF, co morbidities

DETAILED DESCRIPTION:
Study design: A prospective study Sample size: 60 patients (180 readings) Recruitment: Patients will be recruited at the intravitreal injection clinic in Grantham Hospital.

Randomization:

Group 1: control (hypromellose), then Timolol, then Travatan Group 2: Timolol, then Travatan, Hypromellose Group 3: Travatan, then Hypromellose, Timolol

There are three groups of different treatments. Patients recruited will undergone all three groups of treatments. During the first injection visit, patients will be randomized (by envelope method upon recruitment) to start with one of the three groups by envelope method. Treatment given to each group according to randomization in the first visit, then rotated to second and third group at two subsequent injections accordingly.

Injection doctors masked to treatments given.

Study visits:

1. Injection visit

   * Record the anti-VFGF injection to be given
   * Macula disease involved
   * Record no. of previous injections
   * Prophylactic eye drops will be given according to treatment group 1 hour prior injection
   * IOP immediately before injection (without speculum while sitting on table)
   * IOP immediately after injection (without speculum while sitting on table)
   * IOP 30 minutes after injection via iCare
   * Slitlamp examination, document inflammation or complications if any
2. Day 1 follow-up visit

   * IOP via iCare (sitting)
   * Slitlamp examination, document inflammation or complications if any
3. Week 1 follow-up visit

   * IOP via iCare (sitting)
   * Slitlamp examination, document inflammation or complications if any Visit a, b and c will be repeated for 2nd and 3rd injections.

ELIGIBILITY:
Inclusion Criteria:

* AMD patients requiring multiple intravitreal injections (Eylea or Lucentis), not necessarily 3 month loading.
* Age >50
* Chinese patients with ability to read Chinese ICF

Exclusion Criteria:

1. Known glaucoma
2. Corneal disease e.g. corneal scarring or opacity preventing fundal view
3. On steroid or anti glaucoma eye drops
4. Prior vitrectomy or glaucoma surgery
5. Recent intraocular surgery i.e. cataracts surgery
6. Pseudophakic with anterior chamber IOL
7. History of ocular inflammatory disease e.g. uveitis
8. Previous laser iridotomy
9. Recent intravitreal injection of steroid
10. Inability for regular follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
IOP effect of prophylactic IOP lowering eye drops over multiple time points | From baseline to 30 minutes after injection
  IOP in mmHg

SECONDARY OUTCOMES:
IOP effect of intravitreal injection | From baseline to 30 minutes after injection
  IOP in mmHg
IOP response to types of anti VEGF, IOL, type of anti VEGF and co-morbidities | From baseline to 30 minutes after injection
  IOP in mmHg
Inflammation to types of anti VEGF | 1 week post injection
  presence of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- HKSDS Program, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided